CLINICAL TRIAL: NCT05195619
Title: Phase Ib Study to Test the Feasibility and Safety of a Personalized Vaccine in Combination With Low-dose Cyclophosphamide in Patients With Advanced or Metastatic Non Small Cell Lung Cancer (NSCLC)
Brief Title: Personalized DC Vaccines in Non Small Cell Lung Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Dr Hasna Bouchaab, Principal Investigator, Centre Hospitalier Universitaire Vaudois
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHUV-DO-0022-LUNGVAC-2019
Record Dates: First submitted 2021-12-17; First posted 2022-01-19 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Non-small Cell Lung Cancer
Keywords: non-small cell lung cancer; vaccine; cyclophosphamide
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Cyclophosphamide

STUDY DESIGN:
Intervention Model Description: A total of 16 evaluable patients will be recruited, eight in each cohort.
  Cohort 1: metastatic non-small cell lung cancer of any histology without any actionable oncogenic driver treated by SOC. Maintenance treatment with pemetrexed and/or maintenance/continuation of pembrolizumab, nivolumab or atezolizumab is allowed.
  Cohort 2: metastatic NSCLC with actionable oncogenic driver such as EGFR mutation, ROS-1 or ALK rearrangement, currently receiving osimertinib, alectinib, lorlatinib, brigatinib or crizotinib as per SOC in each disease entity.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort 1 (Experimental): metastatic NSCLC of any histology without any actionable oncogenic driver treated by SOC. Maintenance treatment with pemetrexed and/or maintenance/continuation of pembrolizumab, nivolumab or atezolizumab is allowed.
  Interventions: Biological: Autologous dendritic cell vaccine loaded with personalized peptides (PEP-DC vaccine); Drug: Low dose cyclophosphamide
- Cohort 2 (Experimental): metastatic NSCLC with actionable oncogenic driver such as EGFR mutation, ROS-1 or ALK rearrangement, currently receiving osimertinib, alectinib, lorlatinib, brigatinib or crizotinib as per SOC in each disease entity.
  Interventions: Biological: Autologous dendritic cell vaccine loaded with personalized peptides (PEP-DC vaccine); Drug: Low dose cyclophosphamide

INTERVENTIONS:
Biological: Autologous dendritic cell vaccine loaded with personalized peptides (PEP-DC vaccine) — Patients will receive six DC vaccinations Q3W (±3 days) in combination with low dose cyclophosphamide the day before vaccination.
  Each dose of vaccine (PEP-DC) will be split into two injections, which will be administered on W2D2 of each cycle, subcutaneously. Patients will be vaccinated until vaccine exhaustion, disease progression, major toxicity or patient withdrawal, whichever is earlier. Additional DC vaccines may be administered Q3W (±3 days) if available until vaccine exhaustion or disease progression, whichever is earlier.
Drug: Low dose cyclophosphamide — Patients will receive six DC vaccinations Q3W (±3 days) in combination with low dose cyclophosphamide the day before vaccination.

SUMMARY:
Phase Ib clinical trial using autologous dendritric cell (DC) vaccine loaded with personalized peptides (PEP) given in combination with low-dose cyclophosphamide, as standard of care (SOC) therapy in patients with advanced or recurrent metastatic NSCLC.

DETAILED DESCRIPTION:
This is a Phase Ib, single center study evaluating safety and feasibility of DC vaccine (autologous monocyte-derived dendritic cells [moDCs] pulsed with personalized peptides [PEP-DC]) given in combination with low dose cyclophosphamide, as SOC therapy in patients with advanced or recurrent metastatic NSCLC.

Patients with advanced or metastatic NSCLC (metastatic, recurrent and/or unresectable) who received standard of care therapy for advanced disease with no signs of progression will be eligible for this protocol. Patients may have received any number of prior treatments without restriction and any prior immunotherapy before enrollment to the study. However, only patients receiving the maintenance/continuation of SOC treatment options mentioned below are permitted to enter the study. Patients will be enrolled in the following two cohorts:

* Cohort 1: metastatic non-small cell lung cancer of any histology without any actionable oncogenic driver treated by SOC. Maintenance treatment with pemetrexed and/or maintenance/continuation of pembrolizumab, nivolumab or atezolizumab is allowed.
* Cohort 2: metastatic NSCLC with actionable oncogenic driver such as Epidermal Growth Factor Receptors (EGFR) mutation, ROS Proto-Oncogene 1 Receptor Tyrosine Kinase (ROS-1) or anaplastic lymphoma kinase (ALK) rearrangement, currently receiving osimertinib, alectinib, lorlatinib, brigatinib or crizotinib as per SOC in each disease entity.

In both cohorts, patients will receive six DC vaccinations Q3W (±3 days) in combination with low dose cyclophosphamide the day before vaccination. Each dose of vaccine (PEP-DC) will be formulated in two syringes of 525 microL each and administered on week 2 day 2 (W2D2) of each cycle, as subcutaneous injections. Patients will be vaccinated until vaccine exhaustion, disease progression, major toxicity or patient withdrawal, whichever is earlier. Additional DC vaccines may be administered Q3W (±3 days) if available until vaccine exhaustion or disease progression, whichever is earlier.

ELIGIBILITY:
INCLUSION CRITERIA AT SCREENING:

1. Signed informed consent form
2. Histologically confirmed diagnosis of the NSCLC
3. Patients with metastatic, recurrent and/or unresectable NSCLC from stage IIIA (not amenable to radical treatment) to stage IVB provided they have not experienced disease progression on their current standard-of-care therapy at screening, as compared to the tumor assessment at the initiation of standard-of-care therapy as confirmed by Computed tomography/Magnetic Resonance Imaging (CT/MRI).
4. Patients may have received any number of prior treatments without restriction and any prior immunotherapy before enrollment to the study. However, only patients receiving the maintenance/continuation of standard of care (SOC) treatment options mentioned below are permitted to enter the study.
5. Patient may receive only the following maintenance/continuation of SOC therapy during study treatment, as indicated in each case.

   1. Cohort 1: advanced or metastatic non-small cell lung cancer of any histology without any actionable oncogenic driver treated by SOC. Maintenance pemetrexed and/or maintenance pemetrexed + pembrolizumab, pembrolizumab alone, nivolumab, or atezolizumab is allowed.
   2. Cohort 2: advanced or metastatic NSCLC with actionable oncogenic driver such as Epidermal Growth Factor Receptor (EGFR) or anaplastic lymphoma kinase (ALK) or ROS-1-rearrangement, currently receiving osimertinib, alectinib, lorlatinib, brigatinib or crizotinib as per SOC in each disease entity
6. Top 10 personalized peptides (PEP) for the preparation of PEP-DC vaccine has been determined before screening.
7. Patients >18 years of age
8. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
9. Adequate hematologic and end organ function, defined by the following laboratory results obtained within 21 days prior registration:

   * Hemoglobin ≥ 90 g/L
   * Neutrophil count ≥ 1.0 G/L (independently of administration of growth factor within 4 weeks prior registration)
   * Platelet count ≥ 100 G/L
   * Serum creatinine ≤ 1.5x Institutional Upper Limit of Normal (ULN), or Creatinine clearance (CrCl) ≥ 40 mL/min (calculated using the Cockcroft-Gault formula.
   * Serum bilirubin ≤ 1.5 ULN (except subjects with Gilbert's syndrome who must have a total bilirubin level of <3.0 x ULN)
   * Aspartate Aminotransferase/Alanine Aminotransferase (AST/ALT) ≤ 3 x ULN
   * Alkaline phosphatase ≤ 1.5 x ULN
   * Coagulation (INR, PT, aPTT): International Normalized Ratio (INR) or Prothrombin Time (PT) ≤ 1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants; Activated Partial Thromboplastin Time (aPTT) ≤ 1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants.
10. Willing and able to comply with study procedures
11. For women of childbearing potential (WOCBP: sexually mature women who have not undergone a hysterectomy, have not been naturally post-menopausal for at least 12 consecutive months or have a serum follicle-stimulating hormone (FSH) < 40 mIU/ml):

    1. Agreement to follow instructions for method(s) of contraception for the couple from screening until 6 months after last vaccine dose, or last cyclophosphamide
    2. WOCBP must have a negative urine pregnancy test within 7 days, before registration. A positive urine test must be confirmed by a serum pregnancy test.

13. For men and their female partners: agreement to follow instructions for method(s) of contraception for the couple from screening until 6 months after last vaccine dose, or last cyclophosphamide

14. Patient is able to undergo leukapheresis

EXCLUSION CRITERIA AT SCREENING:

1. Pregnant or breast-feeding women
2. Other malignancy within 2 years prior study enrollment, except for those treated with surgical intervention as curative intent in remission.
3. Current, recent (within 4 weeks prior registration), or planned participation in an experimental drug study
4. Patients who show signs of progression according to Response Evaluation Criteria In Solid Tumors (RECIST) 1.1 at screening
5. Planned SOC therapy other than the following:

   * Cohort 1: Maintenance pemetrexed and/or maintenance pemetrexed + pembrolizumab, pembrolizumab alone, nivolumab or atezolizumab is allowed.
   * Cohort 2: osimertinib, alectinib, lorlatinib, brigatinib or crizotinib
6. Known hypersensitivity to any component of the study treatment
7. Any contraindication for using cyclophosphamide
8. Treatment with systemic immunosuppressive medications within 4 weeks prior vaccination (more than an equivalent of 10mg prednisone per day). Patient who has to receive steroid treatment as premedication before pemetrexed are eligible.
9. Administration of a live, attenuated vaccine within 8 weeks before registration

   • Influenza vaccination should be given during influenza season only (approximately October to March). Patients must not receive live, attenuated influenza vaccine within 4 weeks prior registration or at any time during the study.
10. Positive serology defined by the following laboratory results:

    * Positive test for Human Immunodeficiency Virus (HIV)
    * Patients with active or chronic hepatitis B (defined as having a positive hepatitis B surface antigen [HBsAg] test at screening).

      * Patients with past / resolved Hepatitis B Virus (HBV) infection (defined as having a negative HBsAg test and a positive antibody to hepatitis B core antigen [anti-HBc] antibody test) are eligible, if HBV deoxyribonucleic acid (DNA) test is negative.
      * HBV DNA must be obtained in patients with positive hepatitis B core antibody prior start of study treatment.
    * Patients with active hepatitis C. Patients positive for Hepatitis C Virus (HCV) antibody are eligible only if Polymerase Chain Reaction (PCR) is negative for HCV ribonucleic acid (RNA).
11. Severe infections within 8 weeks prior registration including but not limited to hospitalization for complications of infection, bacteremia, or severe pneumonia or signs or symptoms of infection requiring oral or IV antibiotics within 8 weeks prior registration.

    • Patients receiving routine antibiotic prophylaxis (e.g., to prevent chronic obstructive pulmonary disease exacerbation or for dental extraction) are eligible.
12. Any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or render the patient at high risk from treatment complications
13. Treatment with systemic immunostimulatory agents (including but not limited to interferon (IFN)-alpha, interleukin (IL)-2 for any reason within 4 weeks or five half-lives of the drug, whichever is shorter, prior to registration.
14. Treatment with systemic immunosuppressive medications (including but not limited to prednisone, dexamethasone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor [anti-TNF] agents) within 2 weeks prior registration.

    * Patients who are receiving acute, low-dose, systemic immunosuppressant medications (e.g., a one-time dose of dexamethasone for nausea) or physiologic replacement doses (i.e., prednisone 5-7.5 mg/day, or other) for adrenal insufficiency may be enrolled in the study.
    * The use of inhaled corticosteroids and mineralocorticoids (e.g., fludrocortisone) is allowed.

TREATMENT ELIGIBILITY CRITERIA:

Treatment eligibility criteria will be assessed within 14 days before the vaccination period start. Patients are eligible to receive PEP-DC vaccination if they meet all the following criteria:

Key conditions required to initiate vaccination:

1. Confirmation from the CTE GMP laboratory that at least six doses of PEPDC vaccines have been produced and released, and are available for the patient at the CTE GMP facility.
2. Patient does not have any diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding that occurred since enrollment and that give reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that might affect the interpretation of the results or render the patient at high risk from treatment complications.
3. Adequate hematologic and end organ function, defined by the following laboratory results obtained within 2 weeks of first vaccine injection:

   * Hemoglobin ≥ 90 g/L
   * Neutrophil count ≥ 1.0 G/L (independently of administration of growth factor within 4 weeks prior registration)
   * Platelet count ≥ 100 G/L
   * Serum creatinine, ≤ 1.5x Institutional Upper Limit of Normal (ULN), or Creatinine clearance (CrCl) ≥ 40 mL/min (calculated using the Cockcroft-Gault formula.
   * Serum bilirubin ≤ 1.5 ULN (except subjects with Gilbert's syndrome who must have a total bilirubin level of <3.0 x ULN)
   * AST/ALT ≤ 3 x ULN
   * Alkaline phosphatase ≤ 1.5 x ULN
   * Coagulation (INR, PT, aPTT): International Normalized Ratio (INR) or Prothrombin Time (PT) ≤ 1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants; Activated Partial Thromboplastin Time (aPTT) ≤ 1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants.

EXCLUSION CRITERIA FOR VACCINATION:

1. Progression since screening (confirmed by CT scan) according to RECIST 1.1
2. Production of vaccine was not successful (or less than 6 was produced)
3. Treatment with systemic immunosuppressive medications within 4 weeks prior vaccination (more than an equivalent of 10mg prednisone per day) except for premedication given for pemetrexed.
4. Any other diseases, cardiac, metabolic or other dysfunction, physical examination finding or clinical laboratory finding since the screening visit giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or render the patient at high risk from treatment complications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2022-03-22 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Number of patients who receive at least one dose of vaccine | 3.5 years after study activation
  Feasibility will be evaluated by the number of patients who receive at least one dose of vaccine, among all enrolled patients.
Assessment of adverse events | from informed consent form (ICF) signature until 30 days after last injection of DC vaccine/cyclophosphamide
  Safety will be assessed by recording all adverse events (AEs) observed from informed consent form (ICF) signature until 30 days after last injection of DC vaccine/cyclophosphamide.
Assessment of treatment-limiting toxicities | 21 days (i.e. during the full vaccination period)
  Collection of events defined as related to vaccine administration. Patients showing any of them will be withdrawn from the study.

SECONDARY OUTCOMES:
Overall response rate 1 (ORR1) | From enrollment until 6 months
  Rate of patients with objective response (complete response or partial response) across all assessment time-points during the period from enrollment until 6 months.
Overall response rate 2 (ORR2) | From enrollment to progression of the disease (ORR2)
  Rate of patients with objective response (complete response or partial response) across all assessment time-points during the period from enrollment to progression of the disease (ORR2).
Duration of response (DoR) | up to 2 years from 1st vaccine injection
  Defined as the time from objective response (OR) until documented tumor progression date among responders.
Progression-free survival (PFS) | up to 2 years from 1st vaccine injection
  Defined as the time from enrollment until documented tumor progression date (as defined by RECIST v1.1). For patients without progression or death (or patients that withdraw or are lost to follow-up), censoring will occur at the last tumor assessment. PFS rate will be estimated at 6, 12 and 24 months.
Overall survival (OS) | up to 2 years from 1st vaccine injection
  Defined as the time from enrollment until death from any cause. Patients alive at the end of follow-up period will be censored at the last day the patient was known to be alive. OS survival rate will be estimated at 12 and 24 months after the date from first study treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- CHUV Oncology Department, Lausanne, Canton of Vaud, Switzerland